CLINICAL TRIAL: NCT04339764
Title: A Phase I/IIa Trial for Autologous Transplantation of Induced Pluripotent Stem Cell-Derived Retinal Pigment Epithelium for Geographic Atrophy Associated With Age-Related Macular Degeneration
Brief Title: Autologous Transplantation of Induced Pluripotent Stem Cell-Derived Retinal Pigment Epithelium for Geographic Atrophy Associated With Age-Related Macular Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200052; 20-EI-0052
Record Dates: First submitted 2020-04-08; First posted 2020-04-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Dry Age-Related Macular Degeneration; Geographic Atrophy
Keywords: Retina; Cell Therapy; Vitrectomy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving intervention (Experimental): Participants receiving intervention
  Interventions: Drug: iPSC-derived RPE/PLGA transplantation

INTERVENTIONS:
Drug: iPSC-derived RPE/PLGA transplantation — iPSC-derived RPE/PLGA transplantation

SUMMARY:
Background:

Age-related macular degeneration is a common eye disease in people over 50. The "dry" form of the disease can worsen into geographic atrophy, causing blind spots. Researchers want to learn if replacing older eye cells with younger ones can help treat this disease.

Objective:

To test the safety of putting cells inside the eye as a possible future treatment for dry age-related macular degeneration.

Eligibility:

People ages 55 and older who have geographic atrophy with loss of vision. People who have had "wet" macular degeneration in study eye are NOT eligible.

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood and urine tests
* Eye exam
* Eye photos
* Fluorescein angiography. An intravenous (IV) line is placed in an arm vein. A dye is injected. A camera takes pictures of the dye as it flows through the eyes' blood vessels.
* Electroretinography. An electrode is taped to participants' forehead. They sit in the dark. After 30 minutes, numbing eye drops and contact lenses are placed in their eyes. They watch flashing lights.
* Tuberculosis test
* Chest X-ray
* Electrocardiography. Sticky pads are placed on participants' chest to record the heart's electrical activity.

Participants will have at least 14 study visits over 5 and a half years. They will repeat screening tests.

Participants will have retinal pigment epithelium (RPE) transplantation surgery in one eye. For this, cells from participants' blood are turned into RPE cells. These cells are placed in their eye through a cut in their retina. They will get dilating eye drops, an IV line, and anesthesia that may make them sleep. A gas bubble will be put in their eye to help it heal. Participants will receive immunosuppressive medications to avoid transplant rejection.

Participants will be contacted yearly for up to 15 years.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a leading cause of vision loss among the elderly. There are limited treatment options for geographic atrophy (GA), the advanced stage of dry AMD, in which cells of the neurosensory retina and associated retinal pigment epithelium (RPE) gradually degenerate and die. Advances in stem cell biology allowing differentiation of pluripotent cells into RPE in vitro make feasible a cell-based strategy for potential treatment of AMD, and recent methods for induced pluripotent stem cell (iPSC) generation offer promise of individualized autologous therapy. Such an approach involves generation of iPSC from somatic cells taken from a patient with GA, differentiation of iPSC into RPE grown as a monolayer on a thin scaffold in vitro, and transplantation of the RPE/scaffold construct into a small region in the subretinal space of the same patient, with a goal of rescuing the overlying neurosensory retina from further degeneration.

Objective: To evaluate the safety and feasibility of subretinal transplantation of iPSC-derived RPE, grown as a monolayer on a biodegradable poly lactic-co-glycolic acid (PLGA) scaffold, as a potential autologous cell-based therapy for GA associated with AMD.

Study Population: Five participants will undergo RPE transplantation in one eye. Eligible eyes will have GA, best-corrected visual acuity (BCVA) between 20/100 and inclusive of counting fingers (CF), and a fellow eye that has same or better BCVA. If the National Eye Institute (NEI) Data and Safety Monitoring Committee (DSMC) gives clearance to proceed based on review of data from the first cohort, a second cohort of up to seven additional participants with GA, BCVA between 20/80 and CF (inclusive) in the eye being considered for RPE transplantation, and same or better visual acuity in the other eye may undergo the procedure to gather additional safety and potential efficacy data useful for planning future studies. Up to 20 participants may be enrolled to allow for screening failures, for participants withdrawing from the study prior to RPE transplantation, or cases where the RPE cell transplantation does not occur due to intraoperative surgical considerations.

Design: In this phase I/IIa, prospective, single-arm, multi-center clinical trial, participants will undergo subretinal transplantation of autologous iPSC-derived RPE in one eye and will be followed for five years after surgery.

Outcome Measures: The primary outcome measure is the safety of RPE/PLGA transplantation, as determined by assessment of visual acuity change and summary of adverse events at 12 months after RPE/PLGA transplantation. Secondary outcome measures include visual acuity change and adverse event reporting at 24 and 60 months, and changes in the following at 12, 24 and 60 months as compared with baseline, assessed in the transplanted region, and compared where applicable with other areas in the macula, and/or with corresponding regions in the fellow eye: retinal sensitivity and fixation parameters assessed by microperimetry; multifocal electroretinography (mfERG) responses; macular structure on cross-sectional and en face imaging by optical coherence tomography (OCT); macular features on color, single-wavelength reflectance, and fundus autofluorescence (FAF) photography; and fluorescein angiography (FA). Some NEI and JHU participants may undergo imaging of photoreceptor/RPE features using adaptive-optics-assisted macular imaging under a separate NEI protocol (e.g., 15-EI-0020).

ELIGIBILITY:
* INCLUSION CRITERIA:

Participant Eligibility Criteria:

To be eligible, the following inclusion criteria must be met, where applicable.

* Participant must be 55 years of age or older.
* Participant must have a diagnosis of dry AMD, defined as presence (or history, as documented in available color fundus photographs) of at least one medium or large druse (greater than or equal to 63 micrometer diameter) in the macula in at least one eye; AND presence of GA in at least one eye.
* Participant must understand and sign the protocol s informed consent document.
* Any participant of childbearing potential must have a negative pregnancy test at screening and must be willing to undergo pregnancy testing prior to RPE transplantation.
* Any participant of childbearing potential and any participant able to father children who has a partner of childbearing potential must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse, or must agree to practice an effective method of contraception through Month 12 in the study. Acceptable methods of contraception include:

  * Hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
  * Intrauterine device,
  * Barrier methods (diaphragm, condom) with spermicide, or
  * Surgical sterilization (tubal ligation).
* Participant must be medically able to comply with the study treatment (including ability to safely receive anesthesia for surgery), study testing and procedures, and follow-up visits.

Study Eye/Fellow Eye Eligibility Criteria

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below. The fellow eye must also meet the relevant eligibility criteria listed below.

Study Eye Inclusion Criteria:

* The study eye must have one or more regions of geographic atrophy with total area of 1 disc area or more. A region of geographic atrophy is defined as an area of uniform hypofluorescence on fundus autofluorescence (FAF) imaging, with greatest linear dimension at least 500 micrometer, with a border within 500 micrometer of the foveal center, not compatible with pigmentary changes, drusen, RPE detachment, drusenoid RPE detachment, hemorrhage, or other lesion. (Note: If macular geographic atrophy is contiguous with peripapillary atrophy, complicating calculation of total area, only atrophy temporal to a vertical line placed a half disc diameter temporal to the temporal border of the disc will be included in the total area of geographic atrophy calculated for eligibility purposes.)
* For participants in the first cohort, the study eye must have an ETDRS best-corrected visual acuity (BCVA) letter score of <= 53 and >= CF (i.e., Snellen equivalent between 20/100 and CF), and the fellow eye must have a letter score no more than five letters worse than the study eye using Electronic Visual Acuity (EVA) testing. If the study eye is CF vision, then the fellow eye must be both (1) CF or better vision and (2) subjectively as good or better than the study eye according to the subject s perception. (Note: Letter scores within five or fewer letters of each other are accordingly considered equal for eligibility determination, and other factors may be used to select the study eye if both are eligible by BCVA.
* For participants in the second cohort, the study eye must have an ETDRS best-corrected visual acuity (BCVA) letter score of <= 58 and >= CF (i.e., Snellen equivalent between 20/80 and CF), and the fellow eye must have a letter score no more than five letters worse than the study eye using Electronic Visual Acuity (EVA) testing. If the study eye is CF vision, then the fellow eye must be both (1) CF or better vision and (2) subjectively as good or better than the study eye according to the subject s perception. (Note: Letter scores within five or fewer letters of each other are accordingly considered equal for eligibility determination, and other factors may be used to select the study eye if both are eligible by BCVA.
* The compromise in visual acuity for the study eye must be judged predominantly secondary to dry AMD, in the judgment of the investigator.
* The study eye must have clarity of ocular media and degree of pupil dilation sufficient to permit adequate fundus photography and safe vitrectomy surgery.
* The study eye must be either pseudophakic or aphakic.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present:

* Participant is actively receiving another study medication / investigational product (IP).
* Participant has any condition that significantly increases risk of systemic corticosteroids or systemic steroid-sparing immuno-modulatory agents, such as uncontrolled diabetes mellitus, chronic hepatitis or liver failure, chronic renal failure, or present infection with HIV, syphilis, tuberculosis, hepatitis B, or hepatitis C (past infection now resolved, where applicable, is not exclusionary; but persistent infection, even if latent, is exclusionary).
* Participant has diagnosis of a malignancy expected to affect two-year survival.
* Participant is pregnant, breast-feeding, or planning to become pregnant through the first 12 months of the study.
* Participant has a family history of a retinal degeneration other than AMD suspected to play a role in the ocular phenotype of the participant in the judgment of the investigator, based on disease features and mode of inheritance, such as in a case of autosomal dominant retinal degeneration in a parent or child.
* Participant is taking, or has taken within the previous year, medication with known potential toxicity to the retina, optic nerve, or lens (such as chloroquine, hydroxychloroquine, ethambutol).
* Participant is taking any form of systemic anticoagulation which cannot be stopped for an indefinite period of time without significant risk. The determination of significant risk to the participant must be at the discretion of the study investigators and prescribing physician (or qualified alternative).
* Participant is unable or unwilling to give informed consent that includes use of medical records and clinical samples for current and future research.

Study Eye Exclusion Criteria:

* The study eye has macular, subretinal or choroidal neovascularization, as assessed by FA and OCT; or any history of such neovascularization (as assessed by past available records or images).
* The study eye has serous or hemorrhagic pigment epithelial detachment, as assessed by FA and OCT, that is clinically significant in the judgment of the investigator.
* The study eye has a history of photodynamic therapy (PDT) or macular thermal laser photocoagulation, or history of intravitreal injection of anti-vascular endothelial growth factor (VEGF) agents or corticosteroids (excepting medications used peri-operatively at prior cataract surgery). The study eye has had intravitreal injections (anti-complement therapy) for treatment of dry AMD in the previous 12 weeks before enrollment. Any intravitreal injections with anti-complement therapy prior to 12 weeks are not exclusionary.
* The study eye has an axial length > 25.0 mm.
* The study eye has had surgery in the previous 12 weeks, or laser capsulotomy in the previous four weeks.
* The study eye has chronic glaucoma; OR significant ocular hypertension, defined as documented intraocular pressure of >= 26 mmHg on at least two occasions in the absence of self-limited acute glaucoma; OR history of probable or definite steroid response manifesting as acute glaucoma or ocular hypertension, even if self-limited and no longer present; OR the fellow eye has evidence for present or past glaucoma or ocular hypertension judged to significantly impact the risk of glaucoma in the study eye (including history of probable or definite steroid response). (Note: History of self-limited acute glaucoma in a study or fellow eye, if not secondary to steroid response, and if now resolved and not expected to recur (e.g., history of elevated intraocular pressure from retained visco-elastic after cataract surgery), is not exclusionary. History of glaucoma or ocular hypertension in the fellow eye, if not felt to significantly impact risk of glaucoma in the study eye, is not exclusionary.)
* The study eye has a condition materially increasing the risks of surgery or potentially affecting visual function over the next two years in the judgment of the investigator, such as chronic uveitis, diabetic retinopathy, keratitis, scleritis, optic neuropathy, untreated retinal detachment, macular edema from prior vein occlusion or other cause, proliferative vitreoretinopathy (PVR), vitreous hemorrhage, pathologic myopia, etc. A history of such conditions is not exclusionary, if judged to not materially increase risks of surgery or to potentially affect vision in the next two years in the opinion of the investigator.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Summary of adverse events | 12 months compared to final Baseline prior to surgery
  safety measure
Visual acuity change | 12 months compared to final Baseline prior to surgery
  safety measure

SECONDARY OUTCOMES:
Retinal structure (fluorescein angiography) | 12, 24, and 60 month
  Safety and efficacy measure
Retinal Structure (color and autofluorescence imaging) | 12, 24, and 60 months
  Safety and efficacy measure
Multifocal electroretinography responses | 12, 24, and 60 months
  Safety and efficacy measure
Retinal sensitivity and fixation (microperimetry) | 12, 24, and 60 months
  Safety and efficacy measure
Retinal Structure (optical coherence tomography) | 12, 24, and 60 months
  Safety and efficacy measure
Visual acuity change | 24 and 60 months
  Safety and efficacy measure
Summary of adverse events | 24 and 60 months
  Safety and efficacy measure

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-EI-0052.html